CLINICAL TRIAL: NCT03902652
Title: Does Higher (100% Oxygen) Versus Lower (21% Oxygen) During Sustained Inflation and Chest Compression During Cardiopulmonary Resuscitation of Asphyxiated Newborns Improve Time to Return of Spontaneous Circulation - a Randomized Control Trial
Brief Title: Does Higher (100% Oxygen) Versus Lower (21% Oxygen) During CC+SI During CPR of Asphyxiated Newborns Improve Time to ROSC
Acronym: SURV1VE-O2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never commenced at trial site.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00088541
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-06

CONDITIONS: Heart; Arrest, Newborn; Birth Asphyxia; Bradycardia Neonatal
Keywords: Chest Compression; Newborn; Infant; Sustained Inflation
MeSH Terms: conditions — Heart Arrest; Asphyxia Neonatorum | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (21% oxygen during CC+SI) (Experimental): Infants randomized into the "21% oxygen CC+SI group" will receive a SI with a PIP of 25-30 cmH2O while receiving chest compression.
  The SI will be delivered over a period of 20 seconds. This will be followed by PEEP of 5-8 cm water fro 1sec. The use of 20sec SI will be repeated 3 times, which results to 60sec of chest compression. At that time the clinical team will perform an assessment of the newborn's heart rate.
  If heart rate is >60/min continue with standard care as per local hospital policy (standard hospital practice guideline). If heart rate remains <60/min continue with CC+SI for another 20sec at which time a further assessment should be performed. If heart rate remains <60/min continue with CC+SI.
  During CC+SI the clinical team will only use 21% oxygen.
  Interventions: Procedure: Intervention (21% oxygen during CC+SI)
- Intervention (100% oxygen during CC+SI) (Active Comparator): Infants randomized into the "100% oxygen CC+SI group" will receive a SI with a PIP of 25-30 cmH2O while receiving chest compression.
  The SI will be delivered over a period of 20 seconds. This will be followed by PEEP of 5-8 cm water fro 1sec. The use of 20sec SI will be repeated 3 times, which results to 60sec of chest compression. At that time the clinical team will perform an assessment of the newborn's heart rate.
  If heart rate is >60/min continue with standard care as per local hospital policy (standard hospital practice guideline). If heart rate remains <60/min continue with CC+SI for another 20sec at which time a further assessment should be performed. If heart rate remains <60/min continue with CC+SI.
  During CC+SI the clinical team will only use 100% oxygen.
  Interventions: Procedure: Intervention (100% oxygen during CC+SI)

INTERVENTIONS:
Procedure: Intervention (21% oxygen during CC+SI) — Infants randomized into the "21% oxygen CC+SI group" will receive a SI with a PIP of 25-30 cmH2O while receiving chest compression.
  The SI will be delivered over a period of 20 seconds. This will be followed by PEEP of 5-8 cm water fro 1sec. The use of 20sec SI will be repeated 3 times, which results to 60sec of chest compression. At that time the clinical team will perform an assessment of the newborn's heart rate.
  If heart rate is >60/min continue with standard care as per local hospital policy (standard hospital practice guideline). If heart rate remains <60/min continue with CC+SI for another 20sec at which time a further assessment should be performed. If heart rate remains <60/min continue with CC+SI.
  During CC+SI the clinical team will only use 21% oxygen.
  Arms: Intervention (21% oxygen during CC+SI)
Procedure: Intervention (100% oxygen during CC+SI) — Infants randomized into the "100% oxygen CC+SI group" will receive a SI with a PIP of 25-30 cmH2O while receiving chest compression.
  The SI will be delivered over a period of 20 seconds. This will be followed by PEEP of 5-8 cm water fro 1sec. The use of 20sec SI will be repeated 3 times, which results to 60sec of chest compression. At that time the clinical team will perform an assessment of the newborn's heart rate.
  If heart rate is >60/min continue with standard care as per local hospital policy (standard hospital practice guideline). If heart rate remains <60/min continue with CC+SI for another 20sec at which time a further assessment should be performed. If heart rate remains <60/min continue with CC+SI.
  During CC+SI the clinical team will only use 100% oxygen.
  Arms: Intervention (100% oxygen during CC+SI)

SUMMARY:
When newborn babies are born without a heartbeat the clinical team has to provide breathing and chest compressions (what is call cardiopulmonary resuscitation) to the newborn baby. Cardiopulmonary resuscitation is an infrequent event in newborn babies (~1% of all deliveries), approximately one million newborn babies die annually due to lack of oxygen at birth causing being born without a heartbeat. Outcome studies of newborn babies receiving cardiopulmonary resuscitation in the delivery room have reported high rates of death and neurological impairment. This puts a heavy burden on health resources since these infants require frequent hospital re-admission and long-term care.

The poor prognosis raises questions as improve cardiopulmonary resuscitation methods and specifically adapt them to newborn babies to improve outcomes. Currently a 3:1 ratio, which equals 3 chest compressions to one rescue breath to resuscitate a newborn baby. This means that chest compressions are stopped after every 3rd compression to give one rescue breath. The investigators believe that this interruption of chest compressions is bad for the newborn baby and that chest compressions should be continued without interruption while rescue breaths are given continuously. The investigators believe that this approach will allow us to reduce death and long-term burdens in newborn babies born without a heartbeat.

Furthermore, it is not known if rescue breaths given with 100% oxygen or 21% oxygen (room air) is better for newborn babies.

Using continuous chest compressions and rescue breaths without interruptions, this study will compare 21% with 100% oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Term infants requiring chest compressions in the delivery room
* Preterm infants >28 weeks' gestation requiring chest compressions in the delivery room

Exclusion Criteria:

* Infants with congenital abnormality
* Infants with congenital diaphragmatic hernia or congenital heart disease
* Infants who's parents refused to give consent to this study

Ages: 0 Minutes to 20 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-08-27 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Return of spontaneous Circulation | up to 60 Minutes of chest compression
  Duration of chest compression heart rate is >60/min for 60sec.

SECONDARY OUTCOMES:
Mortality | Until infant is discharge from hospital (maximum of 30 weeks after birth)
  Number of infants who die until discharge - comparison between group
Number of Epinephrine dosses during resuscitation | During resuscitation (up to 60 minutes)
  How many doses of epinephrine are given - comparison between group
Rate of brain injury | Until infant is discharge from hospital (maximum of 30 weeks after birth)
  Brain injury either by ultrasound or magnet resonance imaging - comparison between group

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after publication